CLINICAL TRIAL: NCT05265676
Title: A Double-blind, Randomized, Two-period, Two-treatment, Two-sequence, Crossover, Balanced, Single Subcutaneous Dose Pharmacodynamic Comparative Equivalence Study of Enoxaparin Sodium Pre-filled Syringes BP (Injection) 40 mg/0.4 ml (4,000 IU/0.4 mL) of Venus Remedies Limited, India and 'Clexane®' (Enoxaparin Sodium Injection Solution in a Pre-filled Syringe) 4,000 IU (40 mg)/0.4 ml of Sanofi, Germany in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of a Generic Enoxaparin Sodium to Clexane® After Single Subcutaneous Dose in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venus Remedies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C1B00548
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: enoxaparin; low molecular weight heparin; bioequivalence; anticoagulant; antithrombotic; heparin; pharmacodynamic equivalence
MeSH Terms: interventions — enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - AB treatment sequence (Experimental): Period 1 - Test Product (A): Enoxaparin Sodium pre-filled syringe BP 40 mg/0.4 ml of Venus Remedies Limited, India.
  Period 2 - Reference Product (B): 'Clexane®' (Enoxaparin Sodium pre-filled syringe; 40 mg/0.4 ml) of Sanofi, Germany.
  Interventions: Drug: Enoxaparin Sodium (Venus Remedies Limited); Drug: Enoxaparin Sodium (Sanofi)
- Cohort 2 - BA treatment sequence (Experimental): Period 1 - Reference Product (B): 'Clexane®' (Enoxaparin Sodium pre-filled syringe; 40 mg/0.4 ml) of Sanofi, Germany.
  Period 2 - Test Product (A): Enoxaparin Sodium pre-filled syringe BP 40 mg/0.4 ml of Venus Remedies Limited, India.
  Interventions: Drug: Enoxaparin Sodium (Venus Remedies Limited); Drug: Enoxaparin Sodium (Sanofi)

INTERVENTIONS:
Drug: Enoxaparin Sodium (Venus Remedies Limited) — The test drug is enoxaparin sodium pre-filled syringe 40 mg/0.4mL of Venus Remedies Limited, India
  Other Names: Cloti-Xa
Drug: Enoxaparin Sodium (Sanofi) — The reference drug is enoxaparin sodium pre-filled syringe 40 mg/0.4mL of Sanofi, Germany
  Other Names: Clexane

SUMMARY:
This is a single-dose, randomized, double-blind, two-period, two-treatment, two-sequence, crossover, balanced, pharmacodynamic (PD) study with 7 days wash-out period. The objective of this study is to assess the bioequivalence between the Enoxaparin (Venus Remedies Limited, India) and its innovator product (Clexane®, Sanofi, Germany).

DETAILED DESCRIPTION:
Enoxaparin is a widely used low-molecular-weight heparin (LMWH) obtained by alkaline β-eliminative cleavage of heparin benzyl ester derived from the porcine intestinal mucosa. Currently, several biosimilars/generics of LMWHs with differing potencies are being developed and marketed in various parts of the world. They differ in their PK and PD properties, which could be possibly due to the depolymerization processes or the manufacturing methods that result in its structural variability. Therefore, it is important that the potency of each biosimilar LMWH be compared with its innovator's molecule.

The PK properties and bioavailability of LMWHs are routinely determined by pharmacodynamic (PD) surrogates such as Anti-Xa activity, Anti-IIa activity, tissue factor pathway inhibitor (TFPI) and activated partial thromboplastin time (aPTT).

This study was designed as a double-blind, randomized, two-period, two-treatment, two-sequence, crossover, balanced, single-dose pharmacodynamic study in healthy, adult, human subjects under fasting conditions to compare and evaluate the pharmacodynamic profile of test product [Enoxaparin Sodium prefilled syringe BP; 40 mg/0.4 mL (Venus Remedies Limited, India)] with that of reference product ['Clexane®' Enoxaparin Sodium prefilled syringe; 40 mg/0.4 mL (Sanofi, Germany)]. The study was conducted with 24 subjects in accordance with protocol.

After overnight fasting of at least 08 hours, a single dose of either test product or reference product was administered to the subjects slowly by subcutaneous route (shaved abdominal wall) alternated in both period between left or right anterolaterally in a supine posture under the supervision of trained study personnel.

The subjects received the test product (A) and reference product (B) in the study as per the randomization schedule. Participants were randomly selected for one of the two sequences: either AB or BA. The washout period between administration of study drugs in each period was 7 days. Blood samples to assess PD parameters were collected in both study periods at the following time points: pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after dosing.

The Anti-Xa and Anti-IIa activity was measured by the chromogenic method using commercial reagent kits - STA®-liquid Anti-Xa, Diagnostica Stago and Actichrome® Heparin (Anti-IIa) kit, Biomedica Diagnostics, respectively. TFPI was assessed using Enzyme-Linked Immunosorbent Assay (ELISA) kit (Quantikine® Human TFPI ELISA kit) and aPTT was determined using clotting assay reagent kit - STA-C.K. Prest® 5-Diagnostica Stago.

Statistical analysis was performed on the pharmacodynamic data to assess bioequivalence between the test product to the reference product. The average bioequivalence of the products was concluded if two-sided 90% CI for the test to the reference ratio of the population means was within 80% and 125% interval for each of the Ln-transformed data, Amax and AUECt for Anti-Xa and Anti-IIa (primary objective).

ELIGIBILITY:
Inclusion Criteria:- Volunteers must fulfill all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified.

1. Age: 18 to 45 years old, both inclusive.
2. Gender: Male and/or non-pregnant, non-lactating female.

   A. Female of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days prior to first dosing day. They must be using an acceptable form of contraception.

   B. For female of childbearing potential, acceptable forms of contraception include the following:

   i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or

   ii. Barrier methods containing or used in conjunction with a spermicidal agent, or

   iii. Surgical sterilization or

   iv. Practicing sexual abstinence throughout the course of the study.

   C. Female will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

   i. Postmenopausal with spontaneous amenorrhea for at least one year, or

   ii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or

   iii. Total hysterectomy and an absence of bleeding for at least 3 months.
3. BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
4. Volunteer with at least 50 kg weight
5. Able to read & understand informed consent document and give written informed consent to participate in the study
6. Non-smokers and non-tobacco users (i.e. having no past history of smoking and tobacco consuming for at least one year prior to study)
7. Non-alcoholic users will be eligible to participate in this study (i.e. having no past history of drinking alcohol for at least one year prior to study).
8. Able to communicate effectively with study personnel.
9. Willing to provide written informed consent to participate in the study.
10. All volunteers must be judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which will include:

    1. A physical examination (clinical examination) with no clinically significant finding.
    2. Results within normal limits or clinically non-significant for the following tests: haematology, biochemistry, serology, coagulogram and urinalysis

Exclusion Criteria:-

Volunteers must not be enrolled in the study if they meet any one of the following criteria:

1. History of hypersensitivity or idiosyncratic reaction to Enoxaparin Sodium, pork, heparin or its derivatives, other low molecular weight heparins or other related drugs, or any of its formulation ingredients.
2. Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG, chest X-ray recording, obstetrics and gynecological history and examination (for female volunteers)].
3. Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoeitic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
4. History or presence of bronchial asthma.
5. Use of any hormone replacement therapy within 3 months prior to the first dose of study medication.
6. A depot injection or implant of any drug within 3 months prior to the first dose of study medication.
7. Use of CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see http://medicine.iupui.edu/clinpharm/ddis/main-table).
8. History or evidence of drug dependence.
9. History of difficulty with donating blood or difficulty in accessibility of veins.
10. A positive hepatitis screen (includes subtypes B & C).
11. A positive test result for HIV antibody and / or syphilis (RPR).
12. Volunteers who have received a known investigational or equivalent to this drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
13. Volunteers who have donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever is greater.
14. Intolerance to venipuncture
15. Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
16. Institutionalized volunteers.
17. Use of any prescribed medications within 14 days prior to the first dose of study medication.
18. Use of any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
19. Use of grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
20. Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), recreational drugs within 48 hours prior to the first dose of study medication.
21. Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
22. History or presence of active major bleeding.
23. History or presence of Thrombocytopenia.
24. Volunteer having Platelet count lower than lower limit of normal range during screening.
25. Volunteer having Prothrombin Time and Activated Partial Thromboplastin Time 1.1 times higher than the upper limit of normal range during screening.
26. Volunteer having INR outside of normal range during screening.
27. Presence of minor bleeding episodes such as epistaxis, rectal bleeding and gingival bleeding.
28. Volunteers with history of stomach ulcer/duodenal ulcer/intestinal ulcers.
29. Volunteers have undergone any surgery in recent past.
30. Volunteers with the history of piles and fissure.
31. Volunteer having any tattoo or any other type of scar at site of injection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Amax for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  Maximum measured Anti-Xa and Anti-IIa plasma activity over the time span specified
AUECt for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  The area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method, for Anti-Xa and Anti-IIa

SECONDARY OUTCOMES:
AUECi for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  The area under the activity/concentration-time curve from time 0 extrapolated to infinity, for Anti-Xa and Anti-IIa
Tmax for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  Tmax is the time to Amax for Anti-Xa and Anti-IIa
t1/2 for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  apparent first order terminal elimination half-life for Anti-Xa and Anti-IIa
Kel for Anti-Xa and Anti-IIa | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  The terminal elimination rate constant obtained from the slope of the line, fitted by linear least squares regression, through the terminal points of the log (base e) of the activity versus time plot for these points
Amax for ratio of Anti-Xa/Anti-IIa activity, TFPI (Baseline corrected and baseline uncorrected) and aPTT (Baseline corrected and baseline uncorrected). | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  Maximum activity for ratio of Anti-Xa/Anti-IIa and TFPI over the time span specified; maximum clotting time for aPTT
AUECt for ratio of Anti-Xa/Anti-IIa activity, TFPI (Baseline corrected and baseline uncorrected) and aPTT (Baseline corrected and baseline uncorrected) | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  The area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method, for ratio of Anti-Xa/Anti-IIa activity, TFPI (Baseline corrected and baseline uncorrected) and aPTT (Baseline corrected and baseline uncorrected)
AUECi for ratio of Anti-Xa/Anti-IIa activity and TFPI (Baseline corrected and baseline uncorrected) | pre-dose (0.0 hour) and at 0.5, 1.0, 1.5, 2.0, 2.333, 2.667, 3.0, 3.333, 3.667, 4.0, 4.5, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 hours after drug administration
  AUC0-inf is the area under the activity/concentration-time curve from time 0 extrapolated to infinity, for ratio of Anti-Xa/Anti-IIa activity and TFPI (Baseline corrected and baseline uncorrected)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mayur Soni, Principal Investigator — Cliantha Research Limited, India
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saxena S, Chaudhary M, Chaudhary S, Aggarwal A. Bioequivalence of a biosimilar enoxaparin (Cloti-Xa) and its innovator (Clexane(R) ): A single-dose, randomized, double-blind, two-period, two-treatment, two-sequence, crossover, balanced study in healthy human subjects. Pharmacol Res Perspect. 2022 Aug;10(4):e00979. doi: 10.1002/prp2.979. PMID 35762448